CLINICAL TRIAL: NCT05955950
Title: Gratitude Intervention in Promoting Self-care and Improving Negative Psychological States in Patients With Acute Myocardial Infarction: a Randomized Clinical Trial
Brief Title: Gratitude Intervention in Promoting Self-care in Patients With Myocardial Infarction
Acronym: GReATCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UP 5797/22
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Myocardial Infarction, Acute
Keywords: Psychosocial intervention; positive psychology; mental health; self-care,; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized, parallel clinical trial. The study will use a prospective experimental design with Condition and Time as independent variables. The condition has two levels that correspond to the experimental conditions: (a) Gratitude List (aspects of daily experience that one feels grateful for), (b) Any Event List (events of one's own choosing that impressed the participant during the day, whether positive or negative). Time is a repeated measures variable with three levels corresponding to the measurement times: (a) Pre-test (before the intervention), (b) Post-test (at 2 weeks after of the intervention - visit 1) and (c) ) Follow-up (from baseline to 6 months - visit 2).
Who Masked: Outcomes Assessor
Masking Description: Neither the researcher nor the participants will be blind to the group to which they were allocated. Because the first will give the necessary guidance and the second will have knowledge of the existing groups through the TCLE and at the time they receive the instructions. Blinding will only occur for the research participant (scientific initiation scholarship holder or volunteer) who must carry out the return interviews and the application of the questionnaires soon after the end of the intervention and in the 6-month follow-up.
  Primary outcome: Self-care and negative psychological states Secondary outcomes: Change in behavior (physical activity, diet...) and gratitude.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude List (Experimental): Participants must to write 3-5 words a day for 14 days about aspects of their daily experience that they are grateful for.
  Interventions: Behavioral: Gratitude list
- List of any event (Active Comparator): Participants must to write 3-5 words a day for 14 days about events of your own choosing that impressed the participant during the day, whether positive or negative.
  Interventions: Behavioral: List of any event

INTERVENTIONS:
Behavioral: Gratitude list — Participants must to write 3-5 words a day for 14 days about aspects of their daily experience that they are grateful for.
  Arms: Gratitude List
Behavioral: List of any event — Participants must to write 3-5 words a day for 14 days about events of your own choosing that impressed the participant during the day, whether positive or negative.
  Arms: List of any event

SUMMARY:
Introduction: Positive psychological's constructs have shown a direct effect on adherence to pharmacological treatment, diet, physical activity and general commitment to health, in the same way that negative ones, such as depression, anxiety and stress, are associated with worse cardiovascular outcomes and are prevalent in patients with infarction. Objective: To verify whether a gratitude intervention can improve self-care and improve negative psychological states in patients with recent myocardial infarction. Methods: Randomized, parallel clinical trial. The inclusion criteria will be patients with ST-segment elevation myocardial infarction (STEMI) with less than 12 hours of evolution and undergoing primary percutaneous coronary intervention (pPCI). Participants will respond to the socio-demographic and risk factors questionnaire and self-care (ASA-A), anxiety, depression and stress (DASS-21) and gratitude (QG-6) scales. They will be drawn into the gratitude intervention group or neutral events group according to the randomization list. Patients in the intervention group will be tasked with writing down 3 to 5 situations a day for which they are grateful, for 14 days. Patients in the control group will be asked to write down 3 to 5 situations a day that have impacted them, whether good or bad. Both groups will be reassessed after the intervention and after 6 months. Expected results: It is expected that the intervention group will improve self-care and the feeling of gratitude, modify behaviors and decrease negative affects, while the group without intervention will remain unchanged from the beginning of the study to 6 months.

DETAILED DESCRIPTION:
Study design: Randomized, parallel clinical trial. The study will use a prospective experimental design with Condition and Time as independent variables. The condition has two levels that correspond to the experimental conditions: (a) Gratitude List (aspects of daily experience that one feels grateful for), (b) Any Event List (events of one's own choosing that impressed the participant during the day, whether positive or negative). Time is a repeated measures variable with three levels corresponding to the measurement times: (a) Pre-test (before the intervention), (b) Post-test (at 2 weeks after of the intervention - visit 1) and (c) ) Follow-up (from baseline to 6 months - visit 2).

This follow-up period is based on the previous studies. Patients will be invited to participate in the study during hospitalization for AMI. If they agree to participate, they must sign the Free and Informed Consent Form. They will answer the socio-demographic questionnaire and risk factors and self-care scales (ASA-A), anxiety, depression and stress (DASS-21) and gratitude (QG-6).

Envelopes will be opened after the initial interview. Participants will receive instructions for the intervention. Participants will be asked to allocate 10-20 minutes at the end of the day, before bed, for 14 days, to write the lists, according to their allocation group. Studies involving gratitude interventions generally last for two weeks as already explained.

In each group, participants will make a list of up to five items, evaluating the activities of that day. The instructions for the groups were adapted and translated.

For the intervention group (Gratitude List), the instructions will be:

"During the day, many things happen in our lives, big and small, for which we can be grateful. Think about your day and write down up to five things in your life that you are grateful for."

For the control group (List of any event), the instructions were:

"During the day, there are many events in our lives, big and small, that end up affecting us. Think about your day and write down up to five things in your life that affected you." Patients will receive a small notebook for daily notes, starting on the day of discharge. Upon discharge, text messages will be sent to their cell phones with reminders not to forget to start and continue making lists. At the end of 2 weeks of the intervention, patients will be invited to return for a reassessment interview (visit 1), and again at the end of 6 months (visit 2). A 6-month follow-up will be necessary so that we can assess changes in behavior.

To assess the improvement in self-care, the ASA-A scale will be used. To assess emotional factors, the DASS scale (which assesses anxiety, depression and stress) will be used. To assess gratitude in the face of life events, the QG-6 scale and for physical health, a dedicated questionnaire will be used. All scales will be used before and after.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation myocardial infarction (STEMI) patients
* Undergoing primary percutaneous coronary intervention (pPCI).

Exclusion Criteria:

* Patients in need of ventilatory support;
* Over 75 years of age;
* Delirium or dementia reported by the attending physician.
* Not able to answer the questionnaires.
* Very high depression scores requiring referral to psychological care services

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-11-05 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Changes in self-care scores | From baseline to 15 days and from baseline to 6 months
  Changes in self-care scores assessed from Appraisal of Self-care Agency (ASA)
Changes in negative psychological states | From baseline to 15 days and from baseline to 6 months
  Changes in DASS-21 scores

SECONDARY OUTCOMES:
Changes in gratitude scores | From baseline to 15 days and from baseline to 6 months
  Changes in Gratitude Questionnaire - GQ-6 scores
Behavioral changes (physical activity, diet...) | From baseline to 15 days and from baseline to 6 months
  Changes in modifiable cardiovascular risk factors: cholesterol, triglycerides, smoking cessation, etc.

CONTACTS AND LOCATIONS:
Overall Officials: MARCIA M SCHMIDT, Principal Investigator — Institute of Cardiology of Rio Grande do Sul
Locations (1):
- Marcia Moura Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No